CLINICAL TRIAL: NCT05118165
Title: Influence of Optimization of Preoperative Nutritional Status on Perioperative Period in Cardiac Surgery in Patients With Frailty
Brief Title: Influence of Preoperative Nutritional Status on Perioperative Period in Cardiac Surgery in Patients With Frailty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Ingrida Drigotiene, dr, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SAI; SUT_SAI (Other: LithuanianUHS Kaunas Clinic)
Record Dates: First submitted 2021-09-14; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Malnutrition; Protein; Frail Elderly Syndrome
Keywords: preoperative malnutrition; frailty; cardiac surgery
MeSH Terms: conditions — Kwashiorkor; Frailty | interventions — Dietary Supplements; Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- intervention group (Experimental)
  Interventions: Dietary Supplement: Dietary supplement with protein

INTERVENTIONS:
Dietary Supplement: Dietary supplement with protein — Will be included protein supplements in the preoperative diet.
  Arms: intervention group

SUMMARY:
The aim of the study is to determine whether the optimisation of the preoperative nutritional status affects the course of the perioperative period in patients with frailty.

Subjects: Patients 65 and over years of age with frailty or risk of it, with suboptimal nutritional status who are prescribed to elective cardiac surgery .

Research methods: Edmonton Crispness Scale, a Mini Nutritional Assessment (MNA-SF) test will be used to select subjects. Body composition will be examined by bioelectrical impedance analysis (BIA) to determine the degree of phase angle. Changes in laboratory blood tests will be recorded and evaluated The subjects randomly will be divided into control and study groups.

The diet of the patients in the study group will be optimised by protein supplements before elective heart surgery.

The benefits of optimising nutritional status will be evaluated comparing laboratory blood tests, changes in organ function, adverse outcomes, the need for vasoactive drugs, artificial lung ventilation time and length of hospitalisation between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years of age and older.
* Patients for whom cardiac surgery will be performed on a scheduled basis.
* Patients able to move without the help of others except for an aid: a stick, a walker.
* Patients who speak and understand Lithuanian perfectly.
* Patients who have read the informed consent form and confirmed their consent to participate in the study in writing.

Exclusion Criteria:

* Patiens younger than 65 years.
* No written consent of a person to participate in a biomedical research has been obtained;
* Patients with a history of mental illness or central nervous system disorders that interfere with the perception and proper assessment of their health and the meaning and content of the questionnaire / tasks.
* Patients with amputated lower extremities.
* Patients with hepatic insufficiency, one or more of viral hepatitis.
* It is not possible to perform a qualitative physical examination for other reasons (hearing, vision, etc.)
* Allergy to B vitamins.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2021-11-12 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-07-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative outcomes | up to 2 weeks
  The rate of postoperative complications

IPD SHARING:
Plan to Share IPD: No